CLINICAL TRIAL: NCT01729494
Title: Randomized, Open Label, Multicenter Study of Belatacept-based Early Steroid Withdrawal Regimen With Alemtuzumab or rATG Induction Compared to Tacrolimus-based Early Steroid Withdrawal Regimen With rATG Induction in Renal Transplantation
Brief Title: Belatacept Early Steroid Withdrawal Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, E. Steve Woodle, MD, FACS, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BEST
Record Dates: First submitted 2012-10-10; First posted 2012-11-20 (Estimated); Results first posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2020-08

CONDITIONS: Renal Transplantation
Keywords: belatacept; rabbit antithymocyte globulin; alemtuzumab; corticosteroid withdrawal
MeSH Terms: interventions — Alemtuzumab; thymoglobulin; Abatacept; Tacrolimus; Mycophenolic Acid; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Experimental): Alemtuzumab + belatacept + mycophenolate mofetil /Enteric coated mycophenolate sodium + early cessation of steroids
  Interventions: Drug: Alemtuzumab; Drug: Belatacept; Drug: Mycophenolate mofetil; Drug: early cessation of steroids
- Group B (Experimental): Rabbit antithymocyte globulin + belatacept + mycophenolate mofetil /Enteric coated (EC) mycophenolate sodium + early cessation of steroids
  Interventions: Drug: rabbit antithymocyte globulin; Drug: Belatacept; Drug: Mycophenolate mofetil; Drug: early cessation of steroids
- Group C (Active Comparator): Rabbit antithymocyte globulin + tacrolimus + mycophenolate mofetil /Enteric coated (EC) mycophenolate sodium + early cessation of steroids
  Interventions: Drug: rabbit antithymocyte globulin; Drug: Tacrolimus; Drug: Mycophenolate mofetil; Drug: early cessation of steroids

INTERVENTIONS:
Drug: Alemtuzumab — Alemtuzumab will be dosed on day of transplant (Study Day 1) at dose of 30 mg given intravenously (IV) over a period of 2 hours after induction of anesthesia. Methylprednisolone IV will be administered 30-60 minutes prior to the administration of alemtuzumab.
  Other Names: Campath
  Arms: Group A
Drug: rabbit antithymocyte globulin — Rabbit antithymocyte globulin will be dosed post-operatively at a total cumulative dose of 4.0-6.0mg/kg given by days 5-10 post-transplant. It will be administered by local standards of care with the following recommendations. The initial intravenous intra-operative dose will be administered approximately one hour after the methylprednisolone dose. The first dose will be administered so that approximately 25% of the dose is infused prior to revascularization of the graft. Subsequent doses will be administered over a minimum of 4 hours. Premedication with acetaminophen 650mg p.o. and diphenhydramine 25mg p.o. prior to rabbit antithymocyte globulin dose will be given to reduce the incidence of infusion reactions.
  Other Names: Thymoglobulin
  Arms: Group B; Group C
Drug: Belatacept — Belatacept will be administered via intravenous (IV) infusion according to the FDA approved dosage recommendations. Subjects randomized to belatacept arms will receive the first dose of IV belatacept (10 mg/kg) within 12-24 hours post reperfusion. The second dose will be given between post-transplant days 4 -6 (Study Days 5-7), and then study days 14, 28, 56, and 84 (12 weeks) and then subjects will receive belatacept at the maintenance dose of 5 mg/kg every 4 weeks until completion of the trial at 24 months (104 weeks). Study Day 1 is defined as the day of transplant.
  Other Names: Nulojix
  Arms: Group A; Group B
Drug: Tacrolimus — Tacrolimus will be administered orally twice daily (BID). The recommended total initial dose of tacrolimus is 0.1 mg/kg/day in two divided doses orally. Tacrolimus should be started post-transplant within 48 hours or when serum creatinine drops lower than 4mg/dL, whichever comes first. The initial targeted trough level of tacrolimus will be 8 - 12 ng/mL for Days 1 through 30, with dose reduction to achieve a 12-hour trough target of 5 - 10 ng/mL thereafter.
  Other Names: Prograf, various
  Arms: Group C
Drug: Mycophenolate mofetil — The first dose of mycophenolate mofetil/EC mycophenolate sodium will be administered pre-operatively. Patients receiving mycophenolate mofetil will be dosed 1000 mg twice daily (2000mg/day). Patients receiving EC mycophenolate sodium will be dosed 720 mg twice daily (1440 mg/day). Dose may be increased for African American transplant recipients to mycophenolate mofetil 1500 mg twice daily (3000mg/day) or EC mycophenolate sodium 1080 mg twice daily (2160 mg/day).
  Other Names: Cellcept, various, Myfortic
Drug: early cessation of steroids — Glucocorticoid therapy will be administered as described. Methylprednisolone will be administered on Days 1 through 3. Additional tapering doses of glucocorticoids will continue to be given until Day 5 as below:
  Day 1 (day of transplant): 500mg IV prior to alemtuzumab (Group A) or rabbit antithymocyte globulin (Groups B and C) Day 2: 250mg IV Day 3: 125mg IV Day 4: 80mg p.o. Day 5: 60mg p.o. No further steroids
  Other Names: prednisone, various

SUMMARY:
The study purpose is to determine the safety and efficacy of a belatacept-based immunosuppressive regimen (calcineurin inhibitor free) with alemtuzumab or rabbit antithymocyte globulin (rATG) induction and early glucocorticoid withdrawal (CSWD) and a belatacept-based immunosuppressive regimen with tacrolimus-based regimen with rabbit antithymocyte globulin induction and early glucocorticoid withdrawal in renal transplant recipients.

The hypothesis is that a belatacept-based immunosuppressive regimen with alemtuzumab induction, mycophenolate mofetil (MMF)/mycophenolic acid (MPA), and early glucocorticoid withdrawal (Group A) in renal transplant recipients or Belatacept-based immunosuppressive regimen with rabbit antithymocyte globulin induction, MMF/MPA and early glucocorticoid withdrawal (Group B) will lead to less risk of graft loss, patient death, or reduced renal function at 12 months as compared to a tacrolimus-based immunosuppressive regimen with rabbit antithymocyte globulin, MMF/MPA, and early glucocorticoid withdrawal in renal transplant recipients (Group C).

DETAILED DESCRIPTION:
Renal transplant is the most effective treatment for end-stage renal disease. It provides improved survival and quality of life. Maintenance of a functioning renal transplant mandates lifelong immunosuppressive therapy to prevent immune destruction of the graft. Current immunosuppressive regimens yield 1-year survival rates of 89% for cadaveric and 94% for living-donor grafts. Over time, however, there is progressive loss of both subjects and grafts. Five-year graft survival for cadaveric and living related donor renal transplants is 67% and 80%, respectively.

The most common causes of long-term subject and graft loss in kidney transplant recipients are cardiovascular disease and chronic allograft nephropathy (CAN), respectively. Paradoxically, the principal immunosuppressive therapies for renal transplant, the calcineurin inhibitors (CNIs), cyclosporine (CsA) and tacrolimus, directly contribute to long-term allograft loss and subject death, since they are inherently nephrotoxic and can cause or exacerbate cardiovascular risks including hypertension, hypercholesterolemia, and diabetes mellitus.

There is, therefore, a substantial unmet medical need for new therapies in renal transplant that can provide short-term subject and graft survival comparable to the CNIs without their long-term nephrotoxic, cardiovascular, and metabolic effects. Because belatacept can be administered at the time of engraftment rather than in a delayed fashion, as is frequently necessary with CNIs - especially in those allografts with initial impaired renal function-- it affords immunosuppression in a timely manner. Unlike CNIs, the targeted mechanism of action of belatacept should provide immunosuppression without nephrotoxicity or adverse effects on the cardiovascular/metabolic profile.

Glucocorticoids have been a cornerstone of immunosuppressive therapy for six decades. Although glucocorticoids provide potent suppression of allo-immune responses in humans, their adverse effects including infection, diabetes, weight gain, hypertension, hyperlipidemia, bone disease, dermal thinning, collagen loss in multiple tissues, and cataracts, combined with a lack of available therapeutic monitoring all argue against their continued use in transplantation.

Belatacept represents a potential new treatment option for renal transplant recipients, which addresses the current unmet need for an immunosuppressive treatment that provides short-term outcomes comparable to calcineurin inhibitors (CNIs) with the potential to avoid their renal, cardiovascular, and metabolic toxicities. However, the initial Phase 3 studies exhibited in higher rate of acute rejection and malignancy. The malignancies were associated with recipients who were EBV negative at the time of transplant. All EBV negative patients are precluded from treatment with Belatacept. Due to the limitations of Phase 3 trial designs and the required use of basilixumab induction, it is intuitive that the addition of a potent t cell depleting induction agent may decrease the overall acute rejection rate in patients treated with belatacept.

The current study tests these assumptions with the following immunosuppressive regimens. Group A and B consist of potent T-cell depleting induction agents combined with belatacept. Group C represents the most common immunosuppressive regimen currently utilized in the United States. Each of these regimens include early withdrawal of glucocorticoids along with maintenance mycophenolate mofetil.

Based upon the totality of available evidence, the current study offers a favorable benefit/risk profile to study subjects, and the potential to continue to provide important data for the development of new immunosuppressive regimens that address important unmet needs.

The proposed Phase 4 study is designed to determine whether belatacept, in combination with other immunosuppressive agents (rabbit antithymocyte globulin or alemtuzumab, mycophenolate mofetil/EC mycophenolate sodium), may provide acceptable efficacy and safety in de novo kidney transplant recipients, in a regimen that provides simultaneous CNI freedom and early CSWD.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients > 18 years of age.
2. Patient who is receiving a renal transplant from a living or deceased donor.
3. Female patients of child bearing potential must have a negative urine or serum pregnancy test within the past 48 hours prior to study inclusion.
4. The patient has given written informed consent to participate in the study.

Exclusion Criteria:

1. Patient has previously received an organ transplant other than a kidney.
2. Patient is receiving an human leucocyte antigen (HLA) identical living donor transplant.
3. Patient who is a recipient of a multiple organ transplant.
4. Patient has a most recent cytotoxic panel reactive antibody (PRA) of >25% or calculated PRA of > 50% where multiple moderate level HLA antibodies exist and in the opinion of the PI represents substantial HLA sensitization.
5. Patient with a positive T or B cell crossmatch that is primarily due to HLA antibodies.
6. Patient with a donor specific antibody (DSA) as deemed by the local PI to be associated with significant risk of rejection.
7. Patient has received a blood group (ABO) incompatible donor kidney.
8. The donor and/or donor kidney meet any of the following extended criteria for organ donation (ECD):

   * Donor age >/= 60 years OR
   * Donor age 50-59 years and 1 of the following:

     * Cerebrovascular accident (CVA) + hypertension + serum creatinine (SCr) > 1.5 mg/dL OR
     * CVA + hypertension OR
     * CVA + SCr > 1.5 mg/dL OR
     * Hypertension + SCr > 1.5 mg/dL OR
   * Cold ischemia time (CIT) > 24 hours, donor age > 10 years OR
   * Donation after cardiac death (DCD)
9. Recipients will be receiving a dual or en bloc kidney transplant.
10. Donor anticipated cold ischemia is > 30 hours.
11. Recipient that is seropositive for hepatitis C virus (HCV) with detectable Hepatitis C viral load are excluded. HCV seropositive patients with a negative HCV viral load testing may be included.
12. Recipients who are Hepatitis B core antibody seropositive are eligible if their hepatitis B viral loads are negative. After transplant, their hepatitis B viral loads will be monitored every three months for the first year after transplant. If hepatitis B viral loads become positive, patients will be treated per institutional standard of care.
13. Patients who are Hepatitis B surface antibody seropositive and who receive a kidney from a Hepatitis B core surface antibody positive donor may be included.
14. Recipient or donor is known to be seropositive for human immunodeficiency virus (HIV).
15. Recipient who is seronegative for Epstein Barr virus (EBV).
16. Patient has uncontrolled concomitant infection or any other unstable medical condition that could interfere with the study objectives.
17. Patients with thrombocytopenia (PLT < 75,000/mm3), and/or leucopoenia (WBC < 2,000/mm3), or anemia (hemoglobin < 6 g/dL) prior to study inclusion.
18. Patient is taking or has been taking an investigational drug in the 30 days prior to transplant.
19. Patient who has undergone desensitization therapy within 6 months prior to transplant.
20. Patient has a known hypersensitivity to belatacept, tacrolimus, mycophenolate mofetil, alemtuzumab, rabbit anti-thymocyte globulin, or glucocorticoids.
21. Patient is receiving chronic steroid therapy at the time of transplant.
22. Patients with a history of cancer (other than non-melanoma skin cell cancers cured by local resection) within the last 5 years, unless they have an expected disease free survival of > 95%.
23. Patient is pregnant, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by positive human Chorionic Gonadotropin (hCG) laboratory test.
24. Women of childbearing potential must use reliable contraception simultaneously, unless they are status post bilateral tubal ligation, bilateral oophorectomy, or hysterectomy.
25. Patient has any form of substance abuse, psychiatric disorder or a condition that, in the opinion of the investigator, may invalidate communication with the investigator.
26. Inability to cooperate or communicate with the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. Steve Woodle, MD, Principal Investigator — University of Cincinnati
Locations (8):
- United States (8):
  - California Pacific Medical Center, San Francisco, California
  - University of Colorado Denver, Denver, Colorado
  - Tampa General Hospital, Tampa, Florida
  - University of Illinois Medical Center at Chicago, Chicago, Illinois
  - University of Minnesota, Minneapolis, Minnesota
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - University of Wisconsin-Madison, Madison, Wisconsin

REFERENCES:
- [Derived] Pyatt A, McGowan M, Tanaka R, Miyagawa B, Mizuno T, Shields AR, Christianson A, West-Thielke P, Leone JP, Woodle ES, Kaufman D, Wiseman A, Matas AJ, Vinks AA, Alloway RR. Belatacept Pharmacokinetic Analysis of Belatacept Early Steroid Withdrawal Trial (BEST) to Clinical Outcomes and Compared With Reported BENEFIT and BENEFIT-EXT Pharmacokinetic Analysis. Clin Transplant. 2025 Aug;39(8):e70172. doi: 10.1111/ctr.70172. PMID 40704545
- [Derived] Kaufman DB, Woodle ES, Shields AR, Leone J, Matas A, Wiseman A, West-Thielke P, Sa T, King EC, Alloway RR; BEST Study Group. Belatacept for Simultaneous Calcineurin Inhibitor and Chronic Corticosteroid Immunosuppression Avoidance: Two-Year Results of a Prospective, Randomized Multicenter Trial. Clin J Am Soc Nephrol. 2021 Sep;16(9):1387-1397. doi: 10.2215/CJN.13100820. Epub 2021 Jul 7. PMID 34233921
- [Derived] Castro-Rojas CM, Godarova A, Shi T, Hummel SA, Shields A, Tremblay S, Alloway RR, Jordan MB, Woodle ES, Hildeman DA. mTOR Inhibitor Therapy Diminishes Circulating CD8+ CD28- Effector Memory T Cells and Improves Allograft Inflammation in Belatacept-refractory Renal Allograft Rejection. Transplantation. 2020 May;104(5):1058-1069. doi: 10.1097/TP.0000000000002917. PMID 31415033

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Alemtuzumab + belatacept + mycophenolate mofetil /Enteric coated mycophenolate sodium + early cessation of steroids
  Alemtuzumab: Alemtuzumab will be dosed on day of transplant (Study Day 1) at dose of 30 mg given intravenously (IV) over a period of 2 hours after induction of anesthesia. Methylprednisolone IV will be administered 30-60 minutes prior to the administration of alemtuzumab.
  Belatacept: Belatacept will be administered via intravenous (IV) infusion according to the FDA approved dosage recommendations. Subjects randomized to belatacept arms will receive the first dose of IV belatacept (10 mg/kg) within 12-24 hours post reperfusion. The second dose will be given between post-transplant days 4 -6 (Study Days 5-7), and then study days 14, 28, 56, and 84 (12 weeks) and then subjects will receive belatacept at the maintenance dose of 5 mg/kg every 4 weeks until completion of the trial at 24 months (104 weeks). Study Day 1 is the day of transplant.
- Group B: Rabbit antithymocyte globulin + belatacept + mycophenolate mofetil /Enteric coated (EC) mycophenolate sodium + early cessation of steroids
  rabbit antithymocyte globulin: Rabbit antithymocyte globulin will be dosed post-operatively at a total cumulative dose of 4.0-6.0mg/kg given by days 5-10 post-transplant. It will be administered by local standards of care with the following recommendations. The initial intravenous intra-operative dose will be administered approximately one hour after the methylprednisolone dose. The first dose will be administered so that approximately 25% of the dose is infused prior to revascularization of the graft. Subsequent doses will be administered over a minimum of 4 hours. Premedication with acetaminophen 650mg p.o. and diphenhydramine 25mg p.o. prior to rabbit antithymocyte globulin dose will be given to reduce the incidence of infusion reactions.
  Belatacept: Belatacept is administered via intravenous (IV) infusion according to the FDA label.
- Group C: Rabbit antithymocyte globulin + tacrolimus + mycophenolate mofetil /Enteric coated (EC) mycophenolate sodium + early cessation of steroids
  rabbit antithymocyte globulin: Rabbit antithymocyte globulin will be dosed post-operatively at a total cumulative dose of 4.0-6.0mg/kg given by days 5-10 post-transplant. It will be administered by local standards of care with the following recommendations. The initial intravenous intra-operative dose will be administered approximately one hour after the methylprednisolone dose. The first dose will be administered so that approximately 25% of the dose is infused prior to revascularization of the graft. Subsequent doses will be administered over a minimum of 4 hours. Premedication with acetaminophen 650mg p.o. and diphenhydramine 25mg p.o. prior to rabbit antithymocyte globulin dose will be given to reduce the incidence of infusion reactions.
  Tacrolimus: Tacrolimus will be administered orally twice daily (BID).
Period: Overall Study
Arm/Group | Group A | Group B | Group C
Started | 107 | 104 | 105
Completed | 97 | 93 | 94
Not Completed | 10 | 11 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Total
Number analyzed (Participants) | 107 | 104 | 105 | 316
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (13.1) | 51.6 (11.7) | 51.5 (12.3) | 51.4 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 38 | 36 | 104
  Male | 77 | 66 | 69 | 212
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 1 | 5
  Asian | 5 | 0 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 12 | 11 | 19 | 42
  White | 82 | 88 | 80 | 250
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 3 | 5 | 13
Region of Enrollment [Number; unit: participants]
  United States | 107 | 104 | 105 | 316
# Patients with Pre-existing Donor Specific Antibody (DSA) [Count of Participants; unit: Participants] — Patients who have the presence of a donor specific antibody (DSA) at the time of their transplant (baseline)
  Participants | 1 | 4 | 1 | 6
calculated panel reactive antibody (cPRA) % [Mean (Standard Deviation); unit: percentage] | 4.9 (12.7) | 6.4 (16.4) | 5.9 (15.7) | 5.8 (14.6)
Repeat Transplant [Count of Participants; unit: Participants] | 7 | 2 | 3 | 12
Living related donor [Count of Participants; unit: Participants] | 25 | 25 | 33 | 83
Living unrelated donor [Count of Participants; unit: Participants] | 55 | 53 | 47 | 155
Deceased donor [Count of Participants; unit: Participants] | 27 | 26 | 25 | 78
Pre-emptive transplant [Count of Participants; unit: Participants] | 37 | 27 | 40 | 104
Cytomegalovirus (CMV) High Risk status (D+/R-) [Count of Participants; unit: Participants] | 18 | 21 | 25 | 64
Pre-existing diabetes mellitus [Count of Participants; unit: Participants] | 26 | 33 | 33 | 92

OUTCOME MEASURES:

1. Primary Outcome: # Patients With Composite Endpoint of Experiencing Either Death, Graft Loss, or eGFR < 45ml/Min
Description: Number of Patients that experienced patient Death or Graft Loss or had an estimated GFR (eGFR) (MDRD) < 45 mL/min
Time Frame: 12 months
Population: Intent to treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 107 | 104 | 105
Participants | 9 | 15 | 14

2. Secondary Outcome: # Patients Experiencing a Graft Loss But Not Including Patients Who Died With Functioning Graft (Death-censored Graft Loss)
Description: Number of patient who experienced Graft loss, not including (censored) patients who lost graft due to death
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 107 | 104 | 105
Participants | 0 | 1 | 1

3. Secondary Outcome: # Patients With Composite Endpoint of Either Experiencing Death, Graft Loss, or eGFR < 45ml/Min at 24 Months
Description: Composite Endpoint of number of patients who experienced either patient death, allograft loss, or had an eGFR < 45 ml/min/1.73m2
Time Frame: 24 months
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 107 | 104 | 105
Participants | 11 | 13 | 21

4. Secondary Outcome: eGFR (MRDRD) < 45 ml/Min/1.73m2
Description: Patients with reduced Renal function measured by estimated GFR MDRD < 45 ml/min at 24 months
Time Frame: 24 months
Population: Intent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 107 | 104 | 105
Participants | 9 | 8 | 20

5. Secondary Outcome: Biopsy Proven Acute Rejection
Description: Incidence of all biopsy proven acute rejection whether clinically relevant or clinically silent.
Time Frame: 24 months
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 107 | 104 | 105
Participants | 20 | 26 | 7

6. Secondary Outcome: Biopsy Proven Acute Cellular Rejection
Description: Biopsy proven acute cellular rejection (BPACR)
Time Frame: 24 months
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 107 | 104 | 105
Participants | 14 | 22 | 2

7. Secondary Outcome: Biopsy Proven Acute Antibody Mediated Rejection
Description: Incidence of patients experiencing a Biopsy proven acute antibody mediated rejection (BPAMR)
Time Frame: 24 months
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 107 | 104 | 105
Participants | 2 | 2 | 3

8. Secondary Outcome: Biopsy Proven Mixed Acute Rejection
Description: Incidence of patients experiencing a Biopsy proven acute cellular rejection with either DSA positive or C4d staining positive indicating antibody rejection
Time Frame: 24 months
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 107 | 104 | 105
Participants | 4 | 2 | 2

9. Secondary Outcome: # of Patients Developing Denovo Donor Specific Antibody (DSA) Post-transplant
Description: Number of patients (%) with development of denovo DSA after transplant
Time Frame: 24 months
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 89 | 85 | 84
Participants | 5 | 1 | 5

10. Secondary Outcome: Mean eGFR (MDRD) (ml/Min/1.73m2)
Description: Mean eGFR (MDRD) (ml/min/1.73m2) measured for all patients reaching 2 year endpoint
Time Frame: 24 months
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: ml/min/1.73m2
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 96 | 92 | 97
ml/min/1.73m2 | 65.5 (18.9) | 65.3 (19.3) | 63.4 (19.8)

11. Secondary Outcome: Proteinuria UPC Ratio > 0.8
Description: Number of Patients with a Urine protein/creatinine (UPC) ratio > 0.8
Time Frame: 24 months
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 84 | 85 | 84
Participants | 11 | 5 | 21

12. Secondary Outcome: Patient Death
Description: Number of Patients who experienced death, all causes
Time Frame: 24 months
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 107 | 104 | 105
Participants | 2 | 4 | 1

13. Other Pre Specified Outcome: Requirement of T-cell Depleting Therapy for Biopsy Proven Acute Rejection (BPAR)
Description: Number of patients requiring anti-lymphocyte therapy for the treatment of BPAR rejection
Time Frame: 24 months
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 107 | 104 | 105
Participants | 8 | 15 | 0

14. Other Pre Specified Outcome: New Onset Diabetes After Transplantation (NODAT)
Description: Number of patients developing New Onset Diabetes Mellitus after Transplant by one of 5 definitions; only patients without preexisting diabetes were included
Time Frame: 24 months
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 80 | 71 | 72
Participants | 11 | 5 | 12

15. Other Pre Specified Outcome: Time to First BPAR
Description: Mean Time to first episode of BPAR (days)
Time Frame: 24 months
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 107 | 104 | 105
days | 229 (147.7) | 131.6 (119.6) | 159.6 (219.6)

16. Other Pre Specified Outcome: # Patients Experiencing a First Biopsy-proven ACR With Severity Banff > or = 2a Grade
Description: Number of patients with their First BPACR with a Banff grade >= Banff 2a using the Banff 2007 classification system for biopsy grading. Banff grade 2a and above is considered severe cellular rejection and includes grades of Banff 2a, Banff 2b, and Banff 3.
Time Frame: 24 months
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 107 | 104 | 105
Participants | 5 | 12 | 0

17. Other Pre Specified Outcome: Delayed Graft Function
Description: Number of patients experiencing Delayed graft function (DGF) within first week after transplant. DGF is defined as need for dialysis within the first week after transplant.
Time Frame: 24 months
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 107 | 104 | 105
Participants | 3 | 1 | 5

18. Other Pre Specified Outcome: Leukopenia (WBC < 2000/mm3)
Description: Number of patients developing leukopenia defined as WBC < 2000/mm3
Time Frame: 24 months
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 107 | 104 | 105
Participants | 22 | 14 | 15

19. Other Pre Specified Outcome: Steroid Therapy
Description: Number of patients on treatment with corticosteroids at 2 years
Time Frame: 24 months
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 107 | 104 | 105
Participants | 16 | 14 | 9

20. Other Pre Specified Outcome: Discontinuation of Mycophenolate
Description: Number of patients who were discontinued from mycophenolate treatment at 2 years
Time Frame: 24 months
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 107 | 104 | 105
Participants | 11 | 9 | 13

21. Other Pre Specified Outcome: Discontinuation of Study Treatment (Belatacept or Tacrolimus)
Description: Number of patients who had to Discontinue study treatment (belatacept or tacrolimus) at 2 years
Time Frame: 24 months
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 107 | 104 | 105
Participants | 11 | 9 | 5

ADVERSE EVENTS:
Time Frame: Adverse event data was collected in every patient over a 2 year time period.
Description: The definition used for serious adverse events were the same as the standard definition. The definition for adverse events differed only in that the adverse events that were related to immunosuppression were captured and any adverse events of special interest in the study.
Arm/Group | Group A | Group B | Group C
All-Cause Mortality (participants affected / at risk) | 2/107 | 4/104 | 1/105
Serious Adverse Events (participants affected / at risk) | 58/107 | 66/104 | 62/105
Other Adverse Events (participants affected / at risk) | 91/107 | 90/104 | 92/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=107) | Group B (N=104) | Group C (N=105)
Cardiovascular event (Cardiac disorders) | 1 (1) | 9 (12) | 3 (5)
Infection Requiring Hospitalization (Infections and infestations) | 24 | 24 | 23 — all infections which required for participant to be hospitalized.
Renal dysfunction resulting in hospitalization (Renal and urinary disorders) | 30 (53) | 32 (50) | 28 (40)
Malignancy (Immune system disorders) | 7 | 6 | 7
PTLD (Blood and lymphatic system disorders) | 0 | 1 | 0
Nausea/vomiting or GI requiring hospitalization (Gastrointestinal disorders) | 4 (6) | 7 (10) | 13 (16)
Mental status changes or neurological AE's (Nervous system disorders) | 5 (8) | 0 (0) | 5 (9)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=107) | Group B (N=104) | Group C (N=105)
Hematologic events (Blood and lymphatic system disorders) | 59 | 55 | 60
Leukopenia WBC < 2000/mm3 (Blood and lymphatic system disorders) | 22 | 14 | 15
Anemia (Hg < 7gm/dL) (Blood and lymphatic system disorders) | 2 | 3 | 6
Thrombocytopenia (PLT < 50,000/mm3) (Blood and lymphatic system disorders) | 5 | 2 | 1
Gastrointestinal events (Gastrointestinal disorders) | 32 | 34 | 50
Nephrotoxicity events (Renal and urinary disorders) | 22 | 28 | 37
Neurologic events (Nervous system disorders) | 14 | 14 | 33
Electrolyte/metabolic events (Metabolism and nutrition disorders) | 15 | 21 | 32
Wound healing (Skin and subcutaneous tissue disorders) | 7 | 10 | 9
Musculoskeletal/Bone events (Musculoskeletal and connective tissue disorders) | 2 | 6 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-20): https://cdn.clinicaltrials.gov/large-docs/94/NCT01729494/Prot_SAP_000.pdf